CLINICAL TRIAL: NCT04000035
Title: Health in Work - a Measure for Increased Coping and Work Inclusion - An Analysis of Effect of Preventive Information Given at the Workplace - Part 1: Quantitative Data Collection
Brief Title: Health in Work - a Measure for Increased Coping and Work Inclusion
Acronym: HiAforsk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); Norwegian Labour and Welfare Administration (Other); Helse Nord (Industry)
Responsible Party: Principal Investigator, Anje Höper, MD/PhD, Principal investigator, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018/2262(REK)
Record Dates: First submitted 2019-06-11; First posted 2019-06-27 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal Pain; Mental Health Wellness 1; Work-Related Condition
Keywords: sickness absence; psychosocial work environment
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Health

STUDY DESIGN:
Intervention Model Description: two groups: intervention and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health in work (Experimental): The interdisciplinary Health in work intervention consists of three information sessions over the course of one year, with work place processes in between. In the meetings, structured health information about musculoskeletal- and mental disorders is given and put in the context of working and the specific workplace. It is an integrated intervention where information is given together by both healthcare- and NAV-personnel.
  Interventions: Other: Health and work environment information and processes
- Regular work place measures (Active Comparator): Regular work place measures offered by NAV workplace service. Those are interventions given by NAV personnel without healthcare involvement and can be varying.
  Interventions: Other: Health and work environment information and processes

INTERVENTIONS:
Other: Health and work environment information and processes — see arm/group description

SUMMARY:
Health in work - a measure for increased coping and work participation

-An effect analysis of a health- and work environment intervention at the workplace. Part 1:quantitative data collection

The main objective of this study is to investigate the effect of the workplace intervention in the new Norwegian national programme Health in work (HelseIArbeid) through a pragmatic cluster-randomized study.

The main hypothesis is that this interdisciplinary health and welfare intervention at the workplace reduces sick leave and improves mastering of common health problems more efficiently than a conventional welfare intervention. More specifically, it is hypothesized that the Health in work intervention has a better cost-effectiveness in terms of sick leave, use of health services and coping with common health problems indicated by an increased health-related quality of life.

DETAILED DESCRIPTION:
The main objective of this study is to investigate the effect of the workplace intervention in the new Norwegian national concept Health in work (HelseIArbeid) through a pragmatic cluster-randomized study.

The interdisciplinary Health in work intervention consists of three information sessions over the course of one year, with work place processes in between. In the meetings, structured health information about musculoskeletal- and mental disorders is given and put in the context of working and the specific workplace. This includes possibilities to work despite health impairment, work inclusion measures, and discussion on how these could have an influence on the individual, group, management and organizational level. The process involves the workplaces' entire staff (employers and employees). It is an active process and workplaces are stimulated and expected to continue to work with these topics both between sessions and after the last meeting. The interdisciplinary intervention is carried out in a collaboration of qualified personnel from The Norwegian labour and welfare service (NAV) and qualified health personnel from the hospital department of rehabilitation medicine.

The main hypothesis is that this interdisciplinary health and welfare intervention at the workplace reduces sick leave and improves mastering of common health problems more efficiently than a conventional welfare intervention. Conventional workplace measures are given by personnel of NAV workplace service without specialist healthcare involvement, focusing mainly on work inclusion and psychosocial work environment. There are several types of interventions available and they will be customized to the workplace. This means that the control intervention is not standardized and will be varying according to the workplaces' demands.

Participating workplaces are recruited through NAV's conventional contact with workplaces based on an analysis of the workplaces' needs. In the workplaces or workplace units that are interested in participating in the project, the following will be distributed to all staff- including leaders- through the employers' email-list: Information about the project, the informed consent-form and a link to the first electronic questionnaire (Q1). The electronic questionnaire portal is open to answers for two weeks after the initial email. After this time period, the workplaces are randomized to either Health in work or control intervention. A one year intervention period follows as described above. The questionnaire is repeated 12 months (Q2) and 24 months (Q3) after randomization. Q1-3 include the same questions regarding health complaints, health mastering, health related quality of life, and work environment.

Work participation will be assessed at the unit level by data from the employers' sickness absence registers that include both self- and physician-certified sickness absence. Physician-certified sickness absence at the individual level will be gathered from the National register of sickness absence over a four year period from 2 years before randomization to 2 years after. Individual sickness absence will also be assessed by self-report from the questionnaires, considering the last three months prior to the questionnaire.

Data on healthcare utilization at the individual level will be obtained as self-reported data from the questionnaires, as well as objective data from the national register of control and health service refunds (KUHR database) and the Norwegian Patient Register (NPR). These registers include registrations of visits to general practitioners, emergency clinics, physiotherapists, radiologic- laboratory- and psychology/psychiatry and other specialised healthcare services. The study will use the registers' data on number of consultations and costs related to these.

All stakeholders involved in the interventions (workplaces/workplace units, specialist healthcare service and NAV) will keep records of the time used on the interventions (attendance, preparation, implementation, supplementary work, others). Costs related to the different interventions will be assessed from these reports.

Other outcome measures are based on self-reported questionnaire data including health-related quality of life, self-rated health, psychosocial work environment, subjective health complaints, health anxiety, social support and job satisfaction, described in more detail in the outcome section.

Health-economics analyses will be performed on these data in order to determine the cost-effectiveness in terms of sick leave, use of health services and coping with common health problems indicated by an increased health-related quality of life.

This project has a second part not registered here, gathering qualitative data about the Health in work intervention. This will investigate how the intervention works, what the participants´ impression of the intervention is and how the intervention can best be implemented, considering its planned future nationwide application.

CHANGE FROM 2020: Due to the global pandemic, the study was completely halted for a period of 6 months from mid-March through September 2020. Activity was slowly regained after that, but remained on a lower level than normal, fluctuating with changing infection rates in the region. Due to this, there were delays in both collection of informed-consent forms and allocation of workplace units, and the intervention period was prolonged. Consequently, the time-frame between questionnaires one and two was expanded, in collaboration with the reference group and approved by the steering committee. For units included before March 12th 2020, questionnaire Q2 and Q3 will be delayed by 12 months in order to assure that intervention activities can be carried out. For units included in the second half of 2020 the scheduled delay of questionnaire Q2 and Q3 will be 6 months. Units included in 2021 are expected to follow the one year intervention plan. We will take this into consideration in the final statistical analysis.

ELIGIBILITY:
Inclusion Criteria for workplaces/workplace units:

* minimum 8 employees
* accessible data on sickness absence (both self- and physician-certified) in the workplace/workplace unit for the past two years prior to inclusion

Inclusion Criteria for the individual employees:

* all staff employed > 20% in the participating workplaces/workplace units
* Norwegian-speaking

Exclusion Criteria for workplaces/workplace units:

- ongoing profound reorganisation at the workplace/workplace unit (>20% change of employees within workplace unit)

Exclusion Criteria for the individual employees:

- none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1383 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in overall sickness absence rates (self- and physician-certified) at the workplace (unit level) | Time period 24 months prior to randomization compared to the time period 12-24 months after randomization
  Sickness absence data from workplace-registers; Difference-in-difference analyses of sickness absence within and between intervention and control group (% of planned workdays).
Change in healthcare utilization | Time period 24 months prior to randomization compared to the time period 12-24 months after randomization
  Difference-in-difference analyses of health service refunds from National register of control and health service refunds (KUHR database, Helsedirektoratet) and Norwegian Patient Register (NPR, Helsedirektoratet) within and between intervention and control group.
Change in health-related quality of life (HRQoL) by EQ-5D-5L utility value, including EQ-VAS score | Enrollment (Q1) to 12 months (Q2) and 24 months (Q3) after randomization
  Difference-in-difference analyses of HRQoL within and between intervention and control groups by use of EQ-5D/EQ-VAS.The EuroQol descriptive system EQ-5D-5L describes health along five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Participants rate each dimension along five severity levels from no problems (1) to extreme problems (5).The resulting combination (5 to the power of 5 = 3,125 possible combinations) is attached a utility value based on a national value set on a scale from 1(best health) to a 0(or even lower) for worst health.A Norwegian value set is currently being developed.The EQ-VAS (EuroQol vertical visual analogue scale;0 as worst,100 as best possible score) is an integral part that has to be included when using the EQ-5D questionnaire.It offers important, complementary information on respondents' valuations of their HRQoL that are not necessarily captured by use of the 5 dimensional descriptive part of this instrument.
Health-economic analyses | Time period 24 months prior to randomization through 24 months after randomization
  Cost-effectiveness analysis based on primary outcome 3 and cost-benefit analyses based on primary outcome 1 and 2.
  Comparing the intervention arms in terms of incremental costs based on direct- and indirect costs related to interventions throughout the intervention period.

SECONDARY OUTCOMES:
Change in physician-certified sickness absence rates (individual level) | Time period 24 months prior to randomization compared to the time period 12-24 months after randomization
  Data from the Norwegian national register of sickness absence (NAV sykefraværsregister); Difference-in-difference analyses of individual sickness absence rates within and between intervention and control group. Possible impact of Covid-19 pandemic will be addressed.
Change in self-certified sickness absence rates (individual level) | Enrollment (Q1) to 12 months (Q2) and 24 months (Q3) after randomization
  Data from the questionnaires; Difference-in-difference analyses of self-certified sickness absence rates within and between intervention and control group. Possible impact of Covid-19 pandemic will be addressed.
Change in psychosocial work environment by Demand-Control-Support-Questionnaire score | Enrollment (Q1) to 12 months (Q2) and 24 months (Q3) after randomization
  Demand-Control-Support-Questionnaire, short Swedish version (Theorell et al 1991), 11 items on demand and control, and 6 items on support, each with scores 1-4, subscales for demand, control and support. Low scores indicate low demand, control and support. Difference-in-difference analyses of psychosocial work environment within and between intervention and control group. Possible impact of Covid-19 pandemic will be addressed.
Change in social support from colleagues by NDSS-16 score | Enrollment (Q1) to 12 months (Q2) and 24 months (Q3) after randomization
  Nondirective and Directive support Survey (NDSS-16). 16 items scored 1-5. Subscales for directive support (8 items, scale 8-40) and non-directive support (8 items, scale 8-40), the higher the score the more support. Difference-in-difference analyses of social support from colleagues within and between intervention and control group. Possible impact of Covid-19 pandemic will be addressed.
Change in job satisfaction by GJS score | Enrollment (Q1) to 12 months (Q2) and 24 months (Q3) after randomization
  Global Job Satisfaction (GJS). Quinn and Shepard, 1974, 5 items scores 1-5 and 1-3, highest number indicate best job satisfaction. Difference-in-difference analyses of job satisfaction within and between intervention and control group. Possible impact of Covid-19 pandemic will be addressed.
Change in subjective health complaints by SHC score | Enrollment (Q1) to 12 months (Q2) and 24 months (Q3) after randomization
  Subjective Health Complaints (SHC), Eriksen et al. 1999, 29 items scored with 4 levels from 0 (no complaints) to 3 (serious complaints), total score and subscale for mental complaints and musculoskeletal pain. Difference-in-difference analyses of subjective health complaints within and between intervention and control group. Possible impact of Covid-19 pandemic will be addressed.
Change in health anxiety by Whitheley index score | Enrollment (Q1) to 12 months (Q2) and 24 months (Q3) after randomization; comparison with Tromsø Study 7
  Change in score of the revised version of the Whiteley Index-6 scale (WI-6-R).The WI-6-R includes questions regarding health anxiety covering different dimensions such as self-experienced health concern, frequency and severity of health concerns, influence of media on subjective health concerns and experiencing of health symptoms. Each response is graded on a 0-4 Likert Scale, where "0=not at all" to "4=a great deal", enabling to calculate a product score of maximum 24, a higher value indicating higher level of health anxiety.
  Difference-in-difference analyses of health anxiety within and between intervention and control group. Possible impact of Covid-19 pandemic will be addressed.
Change in Satisfaction of life by SWLS score | Enrollment (Q1) to 12 months (Q2) and 24 months (Q3) after randomization
  Satisfaction of life scale (SWLS). Five items where each has response options ranged from 1 (strongly disagree) to 7 (strongly agree), sum score is calculated. The higher the sum score, the higher is the satisfaction of life. Change in sum score of the first 3 items (the last two are sensitive to age). Difference-in-difference analyses of subjective health complaints within and between intervention and control group. Possible impact of Covid-19 pandemic will be addressed.

CONTACTS AND LOCATIONS:
Overall Officials: Nils Fleten, Phd, Study Director — UiT The artic University of Norway / Norwegian Welfare Service Troms
Locations (1):
- University Hospital of Nothern Norway, Tromsø, Norway

REFERENCES:
- [Background] Hoper AC, Terjesen CL, Fleten N. Comparing the New Interdisciplinary Health in Work Intervention With Conventional Monodisciplinary Welfare Interventions at Norwegian Workplaces: Protocol for a Pragmatic Cluster Randomized Trial. JMIR Res Protoc. 2022 Apr 7;11(4):e36166. doi: 10.2196/36166. PMID 35388792
- [Derived] Terjesen CL, Hoper AC, Farbu EH, Olsen JA, Fleten N. Impact of an intersectoral universal workplace intervention on health related quality of life and wellbeing in a pragmatic cluster randomised trial. Sci Rep. 2025 Jul 29;15(1):27715. doi: 10.1038/s41598-025-12221-1. PMID 40730635